CLINICAL TRIAL: NCT03491384
Title: Novel Approaches to Understanding the Role of Cannabinoids and Inflammation in Anxiety
Brief Title: Anxiety, Inflammation, Stress, and Cannabinoids
Status: Completed | Type: Observational
Sponsor: University of Colorado, Boulder (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, L. Cinnamon Bidwell, Assistant Research Professor, University of Colorado, Boulder
Other Study IDs: R01DA04413
Record Dates: First submitted 2018-02-28; First posted 2018-04-09 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Anxiety; Anxiety Disorders; Anxiety Generalized; Anxiety Chronic; Inflammation; Inflammatory Response
Keywords: anxiety; inflammation; cannabis; marijuana; stress
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder; Inflammation; Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples (including DNA analysis) gut microbiome samples (including microbial DNA analysis)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Cannabis (smoked flower, ingested edible) — Self-Directed Use (ad-libitum)

SUMMARY:
This study investigates whether the anxiolytic effects and anti-inflammatory properties of cannabis vary as a function of the ratio of CBD to THC, with the goal that these effects may shed light on the mixed data linking cannabis use and anxiety. Individuals with mild to moderate anxiety who elect to use cannabis (smoked flower or edible) will complete four weeks of observation. Participants complete cognitive tasks, a substance use history, health questionnaires concerning sleep and physical activity, and a blood draw at four different time points (Baseline, after 2 weeks of cannabis use, and immediately before and after self-administration after 4 weeks of use) with the use of a mobile pharmacology laboratory, which goes to a convenient location for each participant to self-administer their cannabis. Participants are then followed for five months to self-report on cannabis use, anxiety, subjective cognitive functioning, sleep quality, and other mental health symptoms.

DETAILED DESCRIPTION:
Marijuana use is on the rise with the number of adults reporting medical and recreational use doubling in the past decade. Among adult medical marijuana users, 39% report using marijuana for the purposes of self-treating or coping with anxiety. Marijuana is approved for medical use in over half the states and is gaining traction for use as an "off-label" add-on therapy for treatment-resistant anxiety and stress-related disorders. Paradoxically, however, while data suggest that marijuana, in particular ∆9-tetrahydrocannabinol (THC), increases anxiety acutely, cross sectional and longitudinal data suggest associations between marijuana use and lower risk for anxiety disorders.

There is some evidence demonstrating that marijuana use is associated with increases in acute anxiety and anxiety disorders. However, other data suggests that marijuana use may be protective for adolescents at-risk for anxiety and decrease the chances of developing an anxiety disorder during college. This finding is consistent with a growing body of evidence from animal models suggesting that marijuana has anxiolytic and anti-inflammatory properties. Clarifying the anxiolytic effects of specific strains that differ in their cannabinoid composition may explain these discrepant findings. Thus, regardless of whether results support or refute the anxiolytic properties of marijuana, findings from this study fill a critical void and can inform public perception.

The study goal is to understand the anxiolytic effects of cannabinoids, in particular the effects of THC-based strains vs. CBD-based strains vs strains containing both THC and CBD in different ratios (1:0, 1:1, or 0:1) on inflammation, cognitive functioning, and anxiety/negative affect. This design will capitalize on the novel opportunity to examine the effects of real world marijuana strains on key outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Non-users of cannabis must have been a non-user of cannabis for at least six months
* If a user of cannabis, at least one episode of lifetime cannabis use and a desire to use cannabis to cope with anxiety.
* Reports at least mild to moderate anxiety (≥5 on GAD-7)

Exclusion Criteria:

* Seeking treatment for a substance use disorder
* Current use of other drugs (e.g., cocaine, methamphetamine)
* Current use psychotropic or steroid-based medications
* Has an immune-relevant disease (e.g. HIV)
* Daily tobacco user
* Currently pregnant or trying to become pregnant
* In treatment for psychotic disorder, bipolar disorder or major depression disorder with suicidal ideation; or a history with these disorders.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cinnamon Bidwell, PhD, Principal Investigator — University of Colorado, Boulder
Locations (1):
- Center for Innovation and Creativity, Boulder, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin-Willett R, Skrzynski CJ, Bryan AD, Bidwell LC. Effects of Cannabinoids on Emotional States and Alcohol Use Among Underrepresented Groups: Moderation by Perceived Discrimination. Hum Psychopharmacol. 2025 Sep;40(5):e70016. doi: 10.1002/hup.70016. PMID 40916181
- [Derived] Skrzynski CJ, Rosa L, Drake A, Bryan AD, Bidwell LC. Experimental study on cannabis use and affect: Effects on reactivity to and recovery from negative stimuli. J Psychopathol Clin Sci. 2025 Aug;134(6):639-650. doi: 10.1037/abn0001023. Epub 2025 Jun 16. PMID 40522823
- [Derived] Bidwell LC, Martin-Willett R, Skrzynski C, Lisano J, Ortiz Torres M, Giordano G, Hutchison KE, Bryan AD. Acute and Extended Anxiolytic Effects of Cannabidiol in Cannabis Flower: A Quasi-Experimental ad libitum Use Study. Cannabis Cannabinoid Res. 2024 Aug;9(4):1015-1027. doi: 10.1089/can.2023.0187. Epub 2024 Jan 22. PMID 38252547
- See also: OASIS Website, CU Change Lab, University of Colorado-Boulder — https://www.colorado.edu/changelab/oasis

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Use: No use of cannabis
- THC Group: Participants used THC dominant products
- CBD Group: Participants used CBD dominant products
- THC+CBD Group: Participants used products with roughly equivalent proportions of THC and CBD
Period: Overall Study
Arm/Group | Non-Use | THC Group | CBD Group | THC+CBD Group
Started | 44 | 105 | 117 | 95
Completed | 42 | 86 | 92 | 80
Not Completed | 2 | 19 | 25 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Use | THC Group | CBD Group | THC+CBD Group | Total
Number analyzed (Participants) | 42 | 86 | 92 | 80 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (14.4) | 31.3 (11.7) | 29.5 (10.9) | 32.3 (12.5) | 31.6 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 50 | 47 | 45 | 169
  Male | 15 | 36 | 45 | 35 | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 5 | 4 | 20
  Not Hispanic or Latino | 38 | 79 | 87 | 76 | 280
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 86 | 92 | 80 | 300
Anxiety: DASS 21 [Mean (Standard Deviation); unit: units on a scale] — Subscale score range 0-42 Normal 0-6; Mild 7-9; Moderate 10-14; Severe 15-19; Extremely severe 20-42
  units on a scale | 9.38 (7.71) | 10.14 (6.69) | 10.46 (7.29) | 10.14 (6.69) | 10.11 (6.86)

OUTCOME MEASURES:

1. Primary Outcome: Change in Anxiety: Depression Anxiety Stress Scale (DASS21).
Description: The DASS21 is a 21-item scale that measures self-reported change in anxiety, depression, and stress symptoms. Participants are asked to use 4-point severity/frequency scales (higher values indicate greater severity) to rate the extent to which they have experienced each state. Scores for Depression, Anxiety and Stress are calculated by summing the scores for the relevant items. Changes in DASS subscale self-report will be tested in relation to THC and CBD blood levels. For this aim, only the Anxiety subscale was used.
  Anxiety subscale score range 0-42 Normal 0-6; Mild 7-9; Moderate 10-14; Severe 15-19; Extremely severe 20-42
Time Frame: Change from baseline to 4 weeks: Baseline (before 4 weeks of cannabis use) and Post-Administration (after 4 weeks of use and after acute self-administration)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non-Use | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 42 | 86 | 92 | 80
units on a scale
  Baseline | 9.38 (7.71) | 10.1 (6.69) | 10.5 (7.29) | 9.85 (6.31)
  4 Weeks | 6.78 (6.63) | 7.14 (5.57) | 5.39 (4.73) | 6.33 (5.6)

2. Primary Outcome: Change in Inflammation: Circulating Levels of Cytokines (Panel of Inflammatory Markers).
Description: Change in inflammation from before to after cannabis use will be tested in relation to THC and CBD blood levels.
  The sum concentration of the cytokines IL-1a, IL-1b, IL-6, IL-8, IL-12, and TNFα, which are generally regarded as pro-inflammatory, will be utilized.
  The range for these values can be from 0 to infinity. Higher values indicate higher (worse) levels of inflammation.
Time Frame: as for outcome 1
Population: Participants were included in inflammatory marker analyses if they had biomarkers available for both timepoints (baseline and 4 weeks). Thus, sample size here is not the same as sample size for self-report based outcomes.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Non-Use | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 24 | 44 | 52 | 51
pg/mL
  Baseline | 484.38 (1280.36) | 110.41 (152.31) | 294.71 (501.34) | 324.04 (871.24)
  4 Week | 62.95 (88.15) | 125.62 (173.02) | 218.07 (487.29) | 338.05 (949.23)

3. Primary Outcome: Patient Global Impression of Change: Global Impression of Change Scale (PGIC).
Description: Patient Global Impression of Change Scale (PGIC) measures self-reported change on a 1-7 scale (i.e. from 1 (very much worse) to 7 (very much improved) in anxiety. Changes in this measure will be tested in relation to THC and CBD blood levels.
  Scale possible score range 0-7, with higher scores indicating the largest amount of possible change.
Time Frame: This was administered only once, at the 4 week timepoint, asking participants to reflect on how much change they had experienced over the past 4 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Use | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 42 | 86 | 92 | 80
score on a scale | 4.4 (0.93) | 5.07 (0.96) | 5.2 (0.73) | 5.24 (0.93)

4. Secondary Outcome: Cognitive Impairment: NIH Toolbox Cognitive Battery, Flanker Inhibitory Control Attention Task (FICA) and International Shopping List Test (ISLT).
Description: Co-outcomes testing multiple domains of thinking, memory, and perception (NIH Toolbox), cognitive impairment in the domains of immediate and delayed recall (ISLT), attention and inhibitory control (FICA). Cognitive outcomes are measured in standard scores (e.g. Range of >70 to >140 (Mean of 100 and SD of 15) with higher scores indicating better performance) and can be averaged to reflect a Standard score of overall cognitive function.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Use | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 42 | 86 | 92 | 80
score on a scale
  Baseline | 108.753 (1.003) | 107.846 (9.442) | 109.799 (9.453) | 108.218 (0.353)
  4 Weeks | 112.917 (10.676) | 112.451 (9.087) | 114.367 (9.14) | 112.772 (11.357)

5. Secondary Outcome: Self-Reported Affect in the Context of Negative Affect Induction Task
Description: Participants reported levels of negative affect on a novel scale from -50 (worst) to +50 (best) while undergoing a guided rumination to induce negative affect.
Time Frame: Acute change in affect from before the negative affect induction task to post-breathing
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Use | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 41 | 86 | 91 | 80
score on a scale
  Baseline | 34.415 (15.56) | 33.518 (17.097) | 33.966 (14.184) | 33.416 (15.25)
  4 weeks | 34.805 (11.9) | 36.687 (14.649) | 36.193 (14.448) | 36.147 (14.312)

6. Secondary Outcome: Change in Depression: Depression Anxiety Stress Scale (DASS21).
Description: The DASS21 is a 21-item scale that measures self-reported change in anxiety, depression, and stress symptoms. Participants are asked to use 4-point severity/frequency scales (higher values indicate greater severity) to rate the extent to which they have experienced each state. For this aim, only the Depression subscale was used.
  Depression subscale score range 0-21 Normal (0 to 4), Mild (5 to 6), Moderate, (7 to 10), Severe (11 to 13), Extremely Severe (14 and above)
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Use | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 42 | 86 | 92 | 80
score on a scale | 10.095 (8.588) | 9.442 (8.921) | 8.901 (8.333) | 8.425 (9.144)

7. Secondary Outcome: Health and Wellbeing
Description: Self-report measure across primary domains of diet, assessment of sleep quality, and health-related well-being. Each domain was assessed with the following single items:
  Diet: "In general, how healthy is your overall diet? Would you say" (response options 0- excellent; 1- very good; 2- good; 3- fair; 4- poor) Sleep Quality: "During the past 2 weeks, how would you rate your sleep quality overall?" (response options 0- very good; 1- fairly good; 2- fairly bad; 3- very bad") Health Related Wellbeing: "In general, how would you describe your health?" (response options 0- excellent; 1- very good; 2- good; 3- fair; 4- poor)
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non-Use | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 42 | 86 | 92 | 80
units on a scale
  Baseline Self Reported Diet | 1.643 (0.932) | 1.791 (0.883) | 1.857 (0.95) | 1.7750 (0.914)
  4 Week Self Reported Diet | 1.659 (0.825) | 1.741 (0.804) | 1.811 (0.792) | 1.772 (0.784)
  Baseline Sleep Quality | 1.167 (0.696) | 1.221 (0.582) | 1.348 (0.67) | 1.362 (0.68)
  4 Week Sleep Quality | 1.167 (0.537) | 1.14 (0.557) | 1.066 (0.611) | 1.2 (0.582)
  Baseline Health-Related Wellbeing | 1.238 (0.726) | 1.291 (0.81) | 1.217 (0.724) | 1.275 (0.675)
  4 Week Health-Related Wellbeing | 1.463 (0.745) | 1.338 (0.816) | 1.618 (0.711) | 1.614 (0.748)

8. Secondary Outcome: Motor Battery: Balance and Motor Function
Description: Motor control assessed via dynamic sway, proprioception, and finger tapping rate. Motor outcomes can be aggregated via Z-score to reflect a Z-score of overall motor function. We calculated the sum of Motor Battery Balance (Eyes Open, Eyes Closed, and Head Back) z-scores. A score of 0 means a participant's balance is at the mean for the sample. Higher scores (scores greater than 0) correspond to worse balance compared to the sample. Scores lower than 0 indicate better balance compared to the sample.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Non-Use | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 17 | 40 | 43 | 45
z-score
  Baseline sum Motor Battery Balance score | 0.0195 (0.007) | 0.0192 (0.006) | 0.0173 (0.005) | 0.0202 (0.014)
  Change in Balance score at 4 weeks | 0.0214 (0.011) | 0.0201 (0.006) | 0.0182 (0.005) | 0.0195 (0.007)

9. Secondary Outcome: Objective Physical Activity/Exercise
Description: Physical activity via objective daily data on wearable watch as measured by average minutes of moderate to vigorous physical activity (MVPA).
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Non-Use | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 29 | 62 | 67 | 49
minutes | 1711.07 (1055.73) | 1751.97 (1075.78) | 1487.81 (1060.91) | 1712.53 (1114.56)

10. Secondary Outcome: Physical Activity/Exercise
Description: Physical activity via subjective self-report data using the Stanford Leisure-Time Activity Categorical item with 6 item responses (L-CAT; 1-6). Scores are reported as a mean between 1 and 6, larger numbers correspond to higher levels of activity.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Use | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 42 | 86 | 92 | 53
score on a scale
  Baseline scores on L-CAT | 3.476 (1.234) | 3.523 (1.326) | 3.571 (1.367) | 3.612 (1.392)
  Change in scores at 4-weeks on L-CAT | 3.415 (1.224) | 3.5 (1.299) | 3.4 (1.234) | 3.481 (1.357)

11. Secondary Outcome: Change in Stress: Depression Anxiety Stress Scale (DASS21).
Description: The DASS21 is a 21-item scale that measures self-reported change in anxiety, depression, and stress symptoms. Participants are asked to use 4-point severity/frequency scales (higher values indicate greater severity) to rate the extent to which they have experienced each state. For this aim, only the Stress subscale was used.
  Stress subscale score range 0-33 Normal (0 to 14), Mild (15 to 18), Moderate, (19 to 25), Severe (26 to 33)
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Use | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 42 | 86 | 92 | 80
score on a scale | 13.714 (8.572) | 13.023 (7.631) | 12.374 (7.136) | 12.4 (7.99)

12. Other Pre Specified Outcome: Exploratory: Daily Follow-Up Messages
Description: Brief self-report from participants on anxiety and sleep in the past 24 hours. These are all 1-item novel questions in a daily, text based survey. Anxiety and sleep are on a scale of 1-10, with higher numbers being more anxiety or better sleep. Score is an average rating over 30 days.
Time Frame: One survey per day for 30 days (at the start of the 4 week study)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non-Use | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 42 | 85 | 92 | 80
units on a scale
  Anxiety Rating | 3.457 (2.386) | 3.394 (2.102) | 3.51 (2.167) | 3.133 (2.066)
  Sleep Quality Rating | 5.687 (1.785) | 5.72 (1.74) | 5.63 (1.818) | 5.455 (1.773)

13. Other Pre Specified Outcome: Exploratory: Monthly Follow-Up Surveys
Description: Self-report from participants on anxiety (DASS anxiety subscale), sleep (novel sleep quality question ranging from 1-10 and 10 being best sleep), subjective cognitive functioning (perceived cognitive ability from the Functional Assessment of Cancer Therapy-Cognitive Function scale as was already reported in secondary measures- see for full description), and general health health (novel health question as was also reported in secondary measures- see for full description).
Time Frame: 5 months (post-study completion)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Non-Use | THC Group | CBD Group | THC+CBD Group
Number analyzed (Participants) | 40 | 57 | 63 | 53
units on a scale
  Anxiety | 3.246 (3.267) | 3.067 (3.15) | 2.844 (2.974) | 3.216 (3.153)
  Sleep | 6.145 (1.671) | 5.763 (1.79) | 5.837 (1.708) | 5.595 (1.626)
  Subjective Cognitive Impairment | 4.657 (11.058) | 5.756 (10.222) | 4.88 (7.918) | 7.718 (14.185)
  General Health | 1.455 (0.779) | 1.367 (0.893) | 1.606 (0.745) | 1.588 (0.777)

ADVERSE EVENTS:
Time Frame: Participants were monitored from Baseline to 4 weeks.
Description: This study was quasi-observational and minimally invasive.
Arm/Group | Non-Use | THC Group | CBD Group | THC+CBD Group
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/86 | 0/92 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/86 | 0/92 | 0/80
Other Adverse Events (participants affected / at risk) | 0/42 | 0/86 | 0/92 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT03491384/Prot_SAP_000.pdf